CLINICAL TRIAL: NCT01209000
Title: Nephrotic Syndrome Study Network Under the Rare Diseases Clinical Research Network
Brief Title: Nephrotic Syndrome Study Network
Acronym: NEPTUNE
Status: Recruiting | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); The NephCure Foundation (Other)
Responsible Party: Principal Investigator, Matthias Kretzler, Professor, University of Michigan
Other Study IDs: 6801; 1U54DK083912 (NIH); NCT01240564 (obsolete NCT alias)
Record Dates: First submitted 2010-07-29; First posted 2010-09-24 (Estimated); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Minimal Change Disease (MCD); Membranous Nephropathy; Glomerulosclerosis, Focal Segmental
Keywords: Focal and Segmental Glomerulosclerosis; Focal & Segmental Glomerulosclerosis; Focal Segmental Glomerulosclerosis; FSGS; Minimal change disease; MCD; Membranous Nephropathy; MN; Nephrotic Syndrome; Neph Syndrome; NEPTUNE; NephCure; Halpin
MeSH Terms: conditions — Nephrosis, Lipoid; Glomerulonephritis, Membranous; Glomerulosclerosis, Focal Segmental; Macular dystrophy, corneal type 1; Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Renal tissue core (from clinically indicated kidney biopsy procedure) Blood products Urine products DNA/RNA specimens (declining consent does not forego participant eligibility)
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (4):
- FSGS/MCD Cohort (Cohort A): Focal Segmental Glomerulosclerosis/Minimal Change Disease (FSGS/MCD) Cohort
  Participants enrolled in NEPTUNE with a biopsy proven histological diagnosis for FSGS or MCD.
  Eligible participants must be scheduled for a clinically indicated renal biopsy.
  Interventions: Procedure: Kidney Biopsy
- MN Cohort (Cohort A): Membranous Nephropathy (MN) Cohort
  Participants enrolled in NEPTUNE with a biopsy proven histological diagnosis for MN.
  Eligible participants must be scheduled for a clinically indicated renal biopsy.
  Interventions: Procedure: Kidney Biopsy
- Other glomerulopathies cohort: Participants enrolled in NEPTUNE and determined to not have FSGS/MCD or MN will be followed in a third group.
  Eligible participants must be scheduled for a clinically indicated renal biopsy.
  Interventions: Procedure: Kidney Biopsy
- cNEPTUNE (Cohort B): Participants < 19 years of age, with < 30 days exposure to immunosuppression therapy who are not scheduled for renal biopsy.

INTERVENTIONS:
Procedure: Kidney Biopsy — Patients scheduled to undergo a clinically indicated kidney biopsy will be requested to consent to an additional renal core, to be set aside until all clinical care is complete.
  Groups: FSGS/MCD Cohort (Cohort A); MN Cohort (Cohort A); Other glomerulopathies cohort

SUMMARY:
Minimal change disease (MCD), focal segmental glomerulosclerosis (FSGS), and Membranous nephropathy (MN), generate an enormous individual and societal financial burden, accounting for approximately 12% of prevalent end stage renal disease (ESRD) cases (2005) at an annual cost in the US of more than $3 billion. However, the clinical classification of these diseases is widely believed to be inadequate by the scientific community. Given the poor understanding of MCD/FSGS and MN biology, it is not surprising that the available therapies are imperfect. The therapies lack a clear biological basis, and as many families have experienced, they are often not beneficial, and in fact may be significantly toxic. Given these observations, it is essential that research be conducted that address these serious obstacles to effectively caring for patients.

In response to a request for applications by the National Institutes of Health, Office of Rare Diseases (NIH, ORD) for the creation of Rare Disease Clinical Research Consortia, a number of affiliated universities joined together with The NephCure Foundation the NIDDK, the ORDR, and the University of Michigan in collaboration towards the establishment of a Nephrotic Syndrome (NS) Rare Diseases Clinical Research Consortium.

Through this consortium the investigators hope to understand the fundamental biology of these rare diseases and aim to bank long-term observational data and corresponding biological specimens for researchers to access and further enrich.

DETAILED DESCRIPTION:
Idiopathic Nephrotic Syndrome (NS) is a rare disease syndrome responsible for approximately 12% of all causes of end-stage kidney disease (ESRD) and up to 20% of ESRD in children. Treatment strategies for Focal and Segmental Glomerulosclerosis (FSGS), Minimal Change Disease (MCD) and Membranous Nephropathy (MN), the major causes of NS, include high dose prolonged steroid therapy, cyclophosphamide, cyclosporine A, tacrolimus, mycophenolate mofetil and other immunosuppressive agents, which all carry significant side effects. Failure to obtain remission using the current treatment approaches frequently results in progression to ESRD with its associated costs, morbidities, and mortality. In the North American Pediatric Renal Trials and Collaborative Studies (NAPRTCS) registry, half of the pediatric patients with Steroid Resistant Nephrotic Syndrome required renal replacement therapy within two years of being enrolled in the disease registry. FSGS also has a high recurrence rate following kidney transplantation (30-40%) and is the most common recurrent disease leading to allograft loss.

The prevailing classification of Nephrotic Syndrome categorizes patients into FSGS, MCD, and MN, if in the absence of other underlying causes, glomerular histology shows a specific histological pattern. This classification does not adequately predict the heterogeneous natural history of patients with FSGS, MCD, and MN. Major advances in understanding the pathogenesis of FSGS and MCD have come over the last ten years from the identification of several mutated genes responsible for causing Steroid Resistant Nephrotic Syndrome (SRNS) presenting with FSGS or MCD histopathology in humans and model organisms. These functionally distinct genetic disorders can present with indistinguishable FSGS lesions on histology confirming the presence of heterogeneous pathogenic mechanisms under the current histological diagnoses.

The limited understanding of FSGS, MCD, and MN biology in humans has necessitated a descriptive classification system in which heterogeneous disorders are grouped together. This invariably consigns these heterogeneous patients to the same therapeutic approaches, which use blunt immunosuppressive drugs that lack a clear biological basis, are often not beneficial, and are complicated by significant toxicity. The foregoing shortcomings make a strong case that concerted and innovative investigational strategies combining basic science, translational, and clinical methods should be employed to study FSGS, MCD, and MN. It is for these reasons that the Nephrotic Syndrome Study Network is established to conduct clinical and translational research in patients with FSGS/MCD and MN.

ELIGIBILITY:
Cohort A (biopsy cohort) Inclusion Criteria:

Patients presenting with an incipient clinical diagnosis for FSGS/MCD or MN or pediatric participants not previously biopsied, with a clinical diagnosis for FSGS/MCD or MN meeting the following inclusion criteria:

* Documented urinary protein excretion ≥1500 mg/24 hours or spot protein: creatinine ratio equivalent at the time of diagnosis or within 3 months of the screening/eligibility visit.
* Scheduled renal biopsy

Cohort B (non-biopsy, cNEPTUNE) Inclusion Criteria:

* Age <19 years of age
* Initial presentation with <30 days immunosuppression therapy
* Proteinuria/nephrotic

  * UA>2+ and edema OR
  * UA>2+ and serum albumin <3 OR
  * UPC > 2g/g and serum albumin <3

Exclusion Criteria (Cohort A&B):

* Prior solid organ transplant
* A clinical diagnosis of glomerulopathy without diagnostic renal biopsy
* Clinical, serological or histological evidence of systemic lupus erythematosus (SLE) as defined by the ARA criteria. Patients with membranous in combination with SLE will be excluded because this entity is well defined within the International Society of Nephrology/Renal Pathology Society categories of lupus nephritis, and frequently overlaps with other classification categories of SLE nephritis (68)
* Clinical or histological evidence of other renal diseases (Alport, Nail Patella, Diabetic Nephropathy, IgA-nephritis, monoclonal gammopathy (multiple myelomas), genito-urinary malformations with vesico-urethral reflux or renal dysplasia)
* Known systemic disease diagnosis at time of enrollment with a life expectancy less than 6 months
* Unwillingness or inability to give a comprehensive informed consent
* Unwillingness to comply with study procedures and visit schedule
* Institutionalized individuals (e.g., prisoners)

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with signs and symptoms of kidney disease consistent with FSGS, MCD, MN or proteinuric renal disease or pediatric participants not previously biopsied, who present for patient care at participating clinical centers will be eligible for Cohort A (biopsy cohort) study population targeted for enrollment into the NEPTUNE study.
  To establish a cohort of pediatric participants with incident nephrotic syndrome, Cohort B, a non-biopsy cohort has been initiated for Protocol V4.0. This population, <19 years of age, presenting for nephrotic syndrome and less than 30 days of immunosuppression therapy exposure, will also be targeted for enrollment into the cNEPTUNE study.
  Potential participants willing to receive their initial care and subsequent follow-up study visits at one of these sites are welcome to participate.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2010-04; Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Event rate of change in urinary protein excretion and renal function. | 60 months
  Defined as remission, partial remission and non-remission
Rate of change in renal function. | 60 months
  Defined as:
  1. 25 mls/min/1.73m2 reduction in follow-up estimated GFR (using the 4-variable MDRD equation for ages ≥18 years and modified Schwartz for ages <18 years) compared to baseline estimated GFR
  2. 50% decline in follow-up estimated GFR compared to baseline measurement
  3. End stage renal disease defined as estimated GFR ≤10cc/min, initiation of maintenance dialysis or preemptive kidney transplantation.

SECONDARY OUTCOMES:
Quality of Life: | 60 months
  Patient-reported outcome will be assessed using Quality of Life questionnaires at regular intervals as stipulated in the visit calendar using the SF-36, PedsQL and the Patient Reported Outcome Measurement Information System (PROMIS) (in the age-appropriate groups).
Malignancies | 60 months
  Any cancer diagnosis of the skin, hematopoietic system, or solid organ after enrollment in NEPTUNE
Infections, Serious and Systemic | 60 months
  Infections including one of the following:
  1. Documented diagnosis of infection of the skin or subcutaneous tissue (e.g. cellulitis), vascular system, peritoneum, or any vital organ requiring the use of parenteral antibiotics and/or oral antibiotics alone or in combination for a treatment interval of ≥72 hours.
  2. Hospitalization for treatment of infection
Thromboembolic Events | 60 months
  Documented diagnosis of one of the following:
  1. Embolic cerebrovascular accident
  2. Deep venous thrombosis
  3. Renal vein thrombosis or
  4. Pulmonary embolus
Hospitalization | 60 months
  Documented hospital admission, including observation for ≥24 hours.
Emergency Department/ Observation Unit Visit | 60 months
  Documented visit to an emergency department or observation unit that does not lead to hospitalization and is less than 24 hours.
Acute Kidney Injury | 60 months
  Documented diagnosis of acute kidney injury as defined by the AKIN (Mehta et al., Critical Care 2007, 11:R31) and/or renal failure requiring renal replacement therapy <3 months.
Death | 60 months
  1. Documentation of death that is secondary to infection or sepsis.
  2. Cardiovascular/Cerebrovascular-related Death: Sudden death; Myocardial infarction; Congestive heart failure; Primary intractable serious arrhythmia; Peripheral vascular disease; Ischemic cerebrovascular accident; Hemorrhagic cerebrovascular accident; Thromboembolic event
  3. Documentation of death secondary to cancer
  4. Other Death: Documentation of death that does not fall into the above categories.
New Onset Diabetes | 60 months
  Diagnosis of diabetes as indicated by 1 or more of the following not present at NEPTUNE Enrollment:
  1. Documented diagnosis of diabetes in medical record
  2. Casual (non-fasting) blood glucose > 200 mg/dL c) Fasting blood glucose > 126 mg/dL d) 2 hour glucose > 200 after oral glucose tolerance test e) chronic use (>6 mos) hypoglycemic therapy outside of pregnancy f) Hemogloblin A1C >= 6.5%

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Kretzler, MD, Principal Investigator — University of Michigan
Locations (44):
- United States (39):
  - University of Southern California-Children's Hospital, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - University of California San Francisco Benioff Children's Hospitals, San Francisco, California
  - Lundquist Biomedical Research Institute at Harbor UCLA Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Anschutz School of Medicine, Aurora, Colorado
  - University of Miami Miller School of Medicine, Miami, Florida
  - Emory University and Children's Healthcare of Atlanta, Atlanta, Georgia
  - John Stroger Cook County Hospital, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Medical Institute, Baltimore, Maryland
  - Kidney Disease Section, NIDDK, NIH, Bethesda, Maryland
  - CS Mott Children's Hospital, University of Michigan, Ann Arbor, Michigan
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University - St Louis, St Louis, Missouri
  - Cohen Children's Hospital, New Hyde Park, New York
  - New York University Medical Center, New York, New York
  - Bellevue Hospital, New York, New York
  - New York University Veterans Administration, New York, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health Levine Children's Hospital, Charlotte, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - University Hospital Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - MetroHealth Hospital at Case Western Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas-Southwestern, Dallas, Texas
  - Texas Children's Hospital - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Providence Medical Research Center, Spokane, Washington
- Canada (5):
  - York Central Hospital, Richmond Hill, Ontario
  - Scarborough Hospital, Scarborough Village, Ontario
  - Credit Valley Hospital, Toronto, Ontario
  - Sunnybrook Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario

REFERENCES:
- [Derived] Wang CS, Troost JP, Wang Y, Greenbaum LA, Gibson K, Trachtman H, Srivastava T, Reidy K, Kaskel F, Sethna CB, Meyers K, Dell KM, Tran CL, Hingorani S, Lemley KV, Lin JJ, Gipson DS. Determinants of medication adherence in childhood nephrotic syndrome and associations of adherence with clinical outcomes. Pediatr Nephrol. 2022 Jul;37(7):1585-1595. doi: 10.1007/s00467-021-05176-8. Epub 2021 Nov 18. PMID 34796395
- [Derived] Solagna F, Tezze C, Lindenmeyer MT, Lu S, Wu G, Liu S, Zhao Y, Mitchell R, Meyer C, Omairi S, Kilic T, Paolini A, Ritvos O, Pasternack A, Matsakas A, Kylies D, Wiesch JSZ, Turner JE, Wanner N, Nair V, Eichinger F, Menon R, Martin IV, Klinkhammer BM, Hoxha E, Cohen CD, Tharaux PL, Boor P, Ostendorf T, Kretzler M, Sandri M, Kretz O, Puelles VG, Patel K, Huber TB. Pro-cachectic factors link experimental and human chronic kidney disease to skeletal muscle wasting programs. J Clin Invest. 2021 Jun 1;131(11):e135821. doi: 10.1172/JCI135821. PMID 34060483
- [Derived] Kang H, Kim DR, Jung YH, Baek CW, Park YH, In Oh J, Kim WJ, Choi GJ. Pre-warming the Streamlined Liner of the Pharynx Airway (SLIPA) improves fitting to the laryngeal structure: a randomized, double-blind study. BMC Anesthesiol. 2015 Nov 20;15:167. doi: 10.1186/s12871-015-0151-4. PMID 26589142
- [Derived] Hogan MC, Lieske JC, Lienczewski CC, Nesbitt LL, Wickman LT, Heyer CM, Harris PC, Ward CJ, Sundsbak JL, Manganelli L, Ju W, Kopp JB, Nelson PJ, Adler SG, Reich HN, Holzmann LB, Kretzler M, Bitzer M. Strategy and rationale for urine collection protocols employed in the NEPTUNE study. BMC Nephrol. 2015 Nov 17;16:190. doi: 10.1186/s12882-015-0185-3. PMID 26577187
- See also: Rare Diseases Clinical Research Networks Homepage — http://rarediseasesnetwork.org
- See also: Patient Advocacy group for FSGS/MCD — http://www.nephcure.org
- See also: Patient advocacy group for MN — http://www.halpinfoundation.org/
- See also: The NEPTUNE Study Homepage — http://www.neptune-study.org